CLINICAL TRIAL: NCT03391310
Title: Use of Honey Versus Standard Treatment for Pressure Ulcers in Critically Ill Children- A Randomized Controlled Trial
Brief Title: Use of Honey for Pressure Ulcers in Critically Ill Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Jhuma Sankar, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110/03.03.2017
Record Dates: First submitted 2017-08-18; First posted 2018-01-05 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Bed Sore; Pressure Ulcer; Pressure Sore; Critically Ill Children
MeSH Terms: conditions — Pressure Ulcer | interventions — Honey

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey dressing group (Experimental): In this group, the wound will be cleaned with normal saline and then honey (medicated ) will be applied to cover the wound surface. The dressing will be changed once soiled (alternate day in most cases). The dressing will be applied for a maximum period upto 8 weeks (in cases of stage IV ulcers) or till healthy granulation tissue appears, whichever is earlier.
  Interventions: Other: Honey (medicated)
- Standard treatment group (No Intervention): In this group, the wound will be first cleaned with 'povidone iodine' and then covered with hydrocolloid dressing changed alternate day for maximum period upto 8 weeks (in cases of stage IV ulcers) or till healthy granulation tissue appears, whichever is earlier.

INTERVENTIONS:
Other: Honey (medicated) — Honey (medicated) dressing will be used in the experimental group
  Other Names: Manuka honey; Leptospermum honey
  Arms: Honey dressing group

SUMMARY:
The enrolled children would be randomized to one of the groups 'study group' or 'Honey dressing group' or 'Group I' (honey dressing containing Active Leptospermum Honey also known as Manuka honey would be used), changed every alternate day for a maximum period of upto 8 weeks (in cases of stage IV ulcers) or till healthy granulation tissue appears, whichever is earlier and 'control group' or 'Standard treatment group ' or 'Group 2' (paraffin gauze is applied after application of povidone iodine). Randomization will be performed as per protocol. Primary outcome will be reduction in time to healing of any stage of pressure ulcer and secondary outcomes will be treatment failure and new onset infection of ulcer.

DETAILED DESCRIPTION:
Children admitted to the PICU would be eligible for inclusion. The interventions will be initiated within the hospital itself. All children will be managed as per standard treatment protocols of the unit for various disease conditions. The enrolled children would be randomized to one of the groups 'study group' or 'Honey dressing group' or 'Group I' (honey dressing containing Active Leptospermum Honey also known as Manuka honey would be used), changed every alternate day for a maximum period of upto 8 weeks (in cases of stage IV ulcers) or till healthy granulation tissue appears, whichever is earlier and 'control group' or 'Standard treatment group ' or 'Group 2' (paraffin gauze is applied after application of povidone iodine). Randomization will be performed as per protocol. Primary outcome will be reduction in time to healing of any stage of pressure ulcer and secondary outcomes will be treatment failure rate and new onset infection of ulcer. The investigators ICU is a fully equipped 8 bedded ICU with all ventilated beds. There are 2 full time consultants, residents and staff with nurse patient ratio of 1:1 to 1:2. Therefore, the investigators are well equipped to treat critically ill children. There will be an in-built mechanism of assuring quality of processes at different steps.

ELIGIBILITY:
Inclusion Criteria:

* All children aged <17 years admitted to the ICU and developing any stage of pressure ulcer due to mechanical pressure or device related pressure during the PICU stay will be eligible for the study

Exclusion Criteria:

Children with pressure ulcers and

* Who are on more than 1 inotrope would be excluded.
* Having signs of acute wound infection,
* Having wounds with > 5 cm diameter,
* Having allergy to honey and not willing to give consent would be excluded.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Time to wound healing | Measured upto 12 weeks of onset of ulcer
  Time to healing of stage 1 to 3 of pressure sore

SECONDARY OUTCOMES:
Rate of new onset infection of the wound | Measured upto 1 week of onset of ulcer
  Wound infection
Rate of treatment failure | Measured upto12 weeks of onset of ulcer
  Wound does not heal
Duration of ICU stay | Measured upto 12 weeks of onset of ulcer
  Length of stay in PICU in days

CONTACTS AND LOCATIONS:
Overall Officials: S K Kabra, MD, Study Chair — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - St. John's Medical College, Bengaluru, Karnataka
  - JIPMER, Puducherry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sankar J, Lalitha AV, Rameshkumar R, Mahadevan S, Kabra SK, Lodha R. Use of Honey Versus Standard Care for Hospital-Acquired Pressure Injury in Critically Ill Children: A Multicenter Randomized Controlled Trial. Pediatr Crit Care Med. 2021 Jun 1;22(6):e349-e362. doi: 10.1097/PCC.0000000000002611. PMID 33181730
- See also: Clinical Trials Registry of India - Registered trial — http://ctri.nic.in/Clinicaltrials/rmaindet.php?trialid=17812&EncHid=25152.16814&modid=1&compid=19